CLINICAL TRIAL: NCT00757302
Title: Evaluation of a New Intraoperative Gamma Camera for the Sentinel Lymph Node Procedure in Breast Cancer
Brief Title: Intraoperative Gamma Camera for Breast Cancer Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut Pluridisciplinaire Hubert Curien. UMR 7178 - CNRS/IN2P3 (Unknown); ULP. F-67037 Strasbourg (Unknown); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4126
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: breast cancer; CarolIReS; intraoperative gamma camera; lymphoscintigraphy; sentinel lymph node; Hundred and ten patients with infiltrative breast cancer or ductal carcinoma in situ (DCIS), diagnosed preoperatively by core biopsy or cytology.
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): For the first 10 patients, only a pre-operative procedure will be performed.
  Interventions: Device: SLN procedure (CarolIReS camera)
- II (Experimental): The last 100 patients will receive the complete procedure.
  Interventions: Device: SLN procedure (CarolIReS camera)

INTERVENTIONS:
Device: SLN procedure (CarolIReS camera) — Group I : The SLN procedure will be initiated 18 hours before surgery using a preoperative injection of colloidal rhenium sulphur and technetium (0.4 ml, 20 MBq of Nanocis®; CIS Bio International, France) at the four cardinal points in the subareolar area. Lymphoscintigraphy will be obtained 3 hours after the injection. Immediately before surgery, the axillary drainage will be checked using the CarolIReS camera (FOV 10x10 cm²).
  Group II : The SLN procedure will be initiated 18 hours before surgery using a preoperative injection of colloidal rhenium sulphur and technetium (0.4 ml, 20 MBq of Nanocis®; CIS Bio International, France) at the four cardinal points in the subareolar area. Lymphoscintigraphy will be obtained 3 hours after the injection. Immediately before surgery, the axillary drainage will be checked using the CarolIReS camera (FOV 10x10 cm²).
  Other Names: gamma camera carolires in detection on sentinel lymph node

SUMMARY:
Aim: This study aims at evaluating the performances of an intraoperative gamma camera (field of view 10X10 cm), named CarolIReS, to detect axillary drainage and to assess the removal of sentinel lymph nodes (SLN) in breast surgery. Patients and Methods: SLN biopsy will be performed on 110 patients and the CarolIReS camera will be used preoperatively to localize SLNs. During surgery, individual removal of SLNs will be performed using a gamma probe named CarolIReS and their activity will be measured with a gamma ray counter. At the end of surgery, the CarolIReS camera will be used again to check the quality of surgery which will be followed by a surgical excision in case of remaining SLNs. Objectives: The main objective of this study is to evaluate the performances of the CarolIReS camera in assessing the axillary drainage of breast tumors and the surgical removal of SLNs. In addition, the possible correlation between the activity, the size, and the metastatic involvement of the SLNs will also be studied.Study hypothesis: Intraoperative cameras could be used to improve the efficiency of the SLN procedure

DETAILED DESCRIPTION:
Group I : The SLN procedure will be initiated 18 hours before surgery using a preoperative injection of colloidal rhenium sulphur and technetium (0.4 ml, 20 MBq of Nanocis®; CIS Bio International, France) at the four cardinal points in the subareolar area. Lymphoscintigraphy will be obtained 3 hours after the injection. Immediately before surgery, the axillary drainage will be checked using the CarolIReS camera (FOV 10x10 cm²). During surgery, the search for radioactive nodes will be performed using the CarolIReS probe. In order to evaluate the CarolIReS camera sensitivity, the activity of the removed SLNs will be measured immediately after their resection by a gamma ray counter and they will then be submitted to pathological analysis with frozen section.

Group II : The SLN procedure will be initiated 18 hours before surgery using a preoperative injection of colloidal rhenium sulphur and technetium (0.4 ml, 20 MBq of Nanocis®; CIS Bio International, France) at the four cardinal points in the subareolar area. Lymphoscintigraphy will be obtained 3 hours after the injection. Immediately before surgery, the axillary drainage will be checked using the CarolIReS camera (FOV 10x10 cm²). During surgery, the search for radioactive nodes will be performed using the CarolIReS probe. In order to evaluate the CarolIReS camera sensitivity, the activity of the removed SLNs will be measured immediately after their resection by a gamma ray counter and they will then be submitted to pathological analysis with frozen section. After SLN removal and during the pathological analysis, the axillary area will once again be checked using the CarolIReS camera (followed by a further surgical excision in the case of remaining SLNs).

When the pathological analysis will diagnose a metastatic SLN, complete axillary lymph node dissection (ALND) will immediately be performed. In the case of negative SLN, serial sections and detection of cytokeratine (AE1/AE3; Dako, Zymed, CA, USA) will be performed during standard pathological analysis. Macrometastases will be defined as clusters of cancer cells ≥2 mm, micrometastases as clusters of cancer cells ≥0.2 mm and <2 mm, and isolated cancer cells as clusters of cancer cells <0.2 mm. ALND will be performed in cases of macro- or micrometastases.

ELIGIBILITY:
Inclusion Criteria:

* Patient major at the time of breast surgery.
* Patient affiliated with a social security.
* Consent dated and signed by the investigator and the subject.
* Subject having been informed of the sentinel lymph node procedure during the visit prior to breast surgery.
* Patient having a unifocal infiltrative breast cancer (less than 2 cm) diagnosed preoperatively by core biopsy or cytology.
* Patient having a ductal carcinoma in situ (DCIS), diagnosed preoperatively by core biopsy or cytology.

Exclusion Criteria:

* Refusal of the patient to be included in the study.
* Pregnant patient or during breastfeeding.
* None of the patients will have undergone chemotherapy, locoregional radiotherapy or prevalent axillary lymph node.
* Diagnosed safeguarding justice and trust.
* Patient with a psychiatric disorder makes it impossible for the collection of informed consent-patient with tumors greater than 2 cm or multifocal.
* Prevalent axillary lymph node.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects for which the gamma camera can detect sentinel lymph nodes (SLN) not identified by other technic. | 1 year

SECONDARY OUTCOMES:
Proportion of subjects with at least one additional sentinel lymph nodes (SLN) detected by preoperative pictures with gamma camera. | 1 year
Proportion of subjects with at least one additional sentinel lymph nodes (SLN) detected by the pictures with gamma camera to intervene. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MATHELIN Carole, MD, Principal Investigator
Locations (1):
- CHRU, Hôpital Civil ,Service de Gynécologie-obstétrique, Strasbourg, France

REFERENCES:
- [Result] Mathelin C, Salvador S, Bekaert V, Croce S, Andriamisandratsoa N, Liegeois P, Prados E, Guyonnet JL, Grucker D, Brasse D. A new intraoperative gamma camera for the sentinel lymph node procedure in breast cancer. Anticancer Res. 2008 Sep-Oct;28(5B):2859-64. PMID 19031925